CLINICAL TRIAL: NCT03621930
Title: REspiratory Syncytial Virus Consortium in EUrope (RESCEU) Study: Defining the Burden of Disease of Respiratory Syncytial Virus in Older Adults in Europe.
Brief Title: RESCEU Study, Defining the Burden of Disease of RSV in Older Adults
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Universiteit Antwerpen (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Louis Bont, Prof. MD, PhD, UMC Utrecht
Other Study IDs: 116019-3
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: RSV Infection; Respiratory Syncytial Virus Infections; Bronchiolitis
Keywords: RESCEU (consortium); RSV; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood:
  * Serum (RSV serology)
  * PaxGene (Transcriptome)
  * Whole blood (cellular immunity, DNA/genome-wide association study (GWAS), epigenetics)
  Swabs:
  * Nasopharyngeal swab (POCT)
  * Nasopharyngeal swab (viral multiplex PCR, deep sequence analysis)
  * Oropharyngeal swab (viral multiplex PCR, deep sequence analysis)
  * Nasopharyngeal swab (microbiome analysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The REspiratory Syncytial virus Consortium in EUrope (RESCEU) is an Innovative Medicine Initiative (IMI) funded by the EU under the H2020 framework to define and understand the burden of disease caused by human respiratory syncytial virus (RSV) infection. RSV causes severe disease in individuals at the extremes of the age spectrum and in high risk groups. It was estimated that RSV was associated with 34 million cases of acute respiratory tract infection (ARTI), 3.4 million ARTI hospitalizations and 55,000 to 199,000 deaths in children <5 years in 2005 worldwide. The estimated burden of disease in older adults is comparable with non-pandemic influenza A (for which a vaccine is available). These estimates were based on limited data and there is a substantial gap in knowledge on morbidity and associated healthcare and social costs in Europe. New vaccines and therapeutics against RSV are in development and could soon be available on the European market. RESCEU will deliver knowledge of the incidence and burden of RSV disease in young children and older adults in Europe, which is essential for stakeholders (governments, etc.) to take decisions about prophylaxis and treatment.

Objective:

To determine the burden of disease due to RSV in older adults.

Study design:

Prospective epidemiological, observational, multi-country, multicenter cohort study.

Study population:

Adults aged 60 years and up (n=1,000) of which approximately 50% is above 75 years of age.

Main study parameters/endpoints:

The primary endpoints of the study are;

* The incidence of RSV infection-associated ARTI.
* RSV associated medically attended (MA) ARTI.
* RSV related hospitalization.

DETAILED DESCRIPTION:
In total, 1000 participants are recruited in three European countries (the Netherlands, Belgium and the United Kingdom). Participants, older adults above the age of 60 years, are recruited from general practitioners offices. Individual participants will be followed for one year (at least one winter season). For the individual participant the study procedures are described below:

Baseline visit:

Baseline visits are performed either at home or at the participating site before the start of the RSV season. The beginning of the season is to be determined per site in accordance to the local virologic surveillance reports. In general, baseline visits are performed between August and the beginning of October.

A questionnaire on demographic, social and clinical status is completed during this visit. Additionally, vital signs are recorded such as oxygen saturation, heart frequency and breathing frequency. During the baseline visit a blood sample (60 ml, serum, paxgene, whole blood) and nasopharyngeal swab (microbiome) will be collected.

Weekly follow-up during the RSV season:

From October until May participants are contacted weekly to check whether there are signs of a respiratory tract infection. If respiratory symptoms are present, the study team will perform a home visit or ask the participant to visit the site to perform a rapid Polymerase Chain Reaction (PCR)-based point of care test (POCT) for RSV using a nasopharyngeal swab. Additionally both an oro- and nasopharyngeal swab are collected for standard PCR, vital signs are recorded. Participants are asked to complete a daily dairy on respiratory symptoms, health care use and quality of life during 28 days from the moment of infection. If symptoms are not present anymore for two consecutive days, the participant can stop completing the diary.

In case of a positive RSV infection, additional sampling is performed by the study team. This consists of a nasopharyngeal swab (microbiome) and blood (Serum/PaxGene/whole blood). The same materials (minus serum and PaxGene sample) are collected again in convalescence (1-2 weeks after infection).

End of season visit:

At the end of the RSV season (May-June), again sampling is performed combined with recording vital signs. Samples collected are; blood (serum/PaxGene) and a nasopharyngeal swab (microbiome). In addition, a questionnaire will completed on respiratory symptoms, health care use, social status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults ≥60 years of age (comorbidity, including chronic heart disease is not an exclusion criterion)
* Willing and able to give written informed consent
* Willing and able to adhere to protocol-specified procedures

Exclusion Criteria:

* Unable to perform the study procedures
* Current alcohol or drug abuse or history of unsuccessfully treated alcohol or drug abuse within the past year
* Dementia
* Life expectancy less than 1 year
* Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination (a more detailed description/list can be found in appendix 3 of the study protocol).
* Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to study participation. The use of topical, inhaled, and nasal glucocorticoids will be permitted (a more detailed description/list can be found in appendix 3 of the study protocol).
* Previous participation in this study or in a RSV interventional trial (vaccine, antivirals).
* Planned leave/holiday during the winter season of more than 1 month in total.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of approximately 1,000 older adults (≥60 years, including approximately 500 ≥75 years). Participants will be randomly recruited from the database of general practitioners in the following countries: the Netherlands (University Medical Centre Utrecht), Belgium (University of Antwerp) and United Kingdom (University of Oxford).
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a Reverse Transcription-Polymerase Chain Reaction (RT-PCR) confirmed RSV infection (incidence of RSV infection). | Data is collected during the RSV season by weekly contact and viral swab diagnostics for RSV in case of respiratory infection. Medically attended RSV will be recorded throughout the one year follow-up.
  The main outcome of the study is to determine the burden of RSV in the older adult population. Therefore the incidence rate of all RSV in the overall study population of older patients is investigated, including medically attended RSV infection-associated ARTI in both inpatients and outpatients. Nasal swabs are collected by the study team in case of a respiratory infection and tested with RT-PCR for presence of RSV. The incidence of RSV is calculated by dividing the number of RSV positive infections by the total number of study participants. The number of RSV positive infections divided by the total number of infections is calculated as well.

SECONDARY OUTCOMES:
The incidence rate of all-cause MA-ARTI or events leading to worsening of cardiorespiratory status (based on questionnaires at baseline and after one year of follow-up). | Data on worsening of cardiorespiratory status is collected during individual study participation of 1 year
  worsening of cardiorespiratory status is monitored using the questionnaire data collected at baseline and follow-up after 1 year. This includes questions on medication usage, new chronic diagnoses and doctor visits for all cause respiratory illness.
RSV-related mortality through the RSV season. | Data on mortality is collected during individual study participation of 1 year
  Mortality through the RSV season. RSV-associated deaths are recorded and verified by the presence of an active infection with PCR proven RSV-infection around the time of death. Data is recorded in questionnaires during and after the winter season and based on hospital case-report forms (CRF's) in case of in-hospital death.
Non-RSV related mortality through the RSV season. | Data on mortality is collected during individual study participation of 1 year
  Mortality through the RSV season. All-cause mortality is recorded. Data is recorded in questionnaires during and after the winter season and based on hospital case-report forms (CRF's) in case of in-hospital death.
Health care costs for RSV-associated ARTI. | Data on health care costs are collected during individual study participation of 1 year
  Health care cost are examined with regard to resource usage such as hospitalization, hospital duration, incidence and duration of intensive care unit stay, supplemental oxygen use, antibiotic and antiviral use and number of outpatient visits (e.g., ER visit, physician office/outpatient visits). The costs of these resource use are calculated to determine the health care cost associated with an RSV infection.
Health care costs for all-cause MA-ARTI. | Data on health care costs are collected during individual study participation of 1 year
  Health care cost for all-cause medically attended ARTI are examined with regard to resource usage such as hospitalization, hospital duration, incidence and duration of intensive care unit stay, supplemental oxygen use, antibiotic and antiviral use and number of outpatient visits (e.g., ER visit, physician office/outpatient visits).The costs of these resource use are calculated to determine the health care cost associated with an RSV infection.
The incidence rate of RSV-associated secondary bacterial pneumonia events | Data on the incidence of pneumonia are collected during individual study participation of 1 year
  defined as pneumonia within 21 days after RSV infection and associated antibiotic use.
Change in frailty over the course of study using the Groningen Frailty indicator (GFI) questionnaire. | Data on the change in frailty is collected during individual study participation of 1 year
  Frailty is assessed using the Groningen Frailty Indicator questionnaire which is included in the baseline and 1 year follow-up questionnaire. The GFI is a 15-item screening instrument to determine the level of frailty, which is available in a professional and self-report version. It measures the loss of functions and resources in 4 domains: physical (mobility functions, multiple health problems, physical fatigue, vision, hearing), cognitive (cognitive dysfunction), social (emotional isolation), and psychological (depressed mood and feelings of anxiety). All answer categories were dichotomized and a score of 1 indicates a problem or dependency. The range of the GFI score is 0 to 15. Geriatric experts agreed that a score of 4 or higher represents moderate to severe frailty
Sample collection for biomarker analysis to investigate possible biomarkers which are predictive of severe or complicated RSV disease in older adults | Samples are collected at various timepoints during the one year study participation.
  Blood sampling (serum/paxgene/whole blood) as well as viral and microbiome sampling using naso-/oropharyngeal swabs is performed to collect biomaterials for biomarker research on RSV severity and susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Louis J Bont, MD, PhD, Principal Investigator — University Medical Centre Utrecht, UMCU
Locations (3):
- University of Antwerp, Antwerp, Antwerpen, Belgium
- University Medical Centre Utrecht, Utrecht, Netherlands
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salaun B, De Smedt J, Vernhes C, Moureau A, Oner D, Bastian AR, Janssens M, Balla-Jhagjhoorsingh S, Aerssens J, Lambert C, Coenen S, Butler CC, Drysdale SB, Wildenbeest JG, Pollard AJ, Openshaw PJM, Bont L. T cells, more than antibodies, may prevent symptoms developing from respiratory syncytial virus infections in older adults. Front Immunol. 2023 Oct 13;14:1260146. doi: 10.3389/fimmu.2023.1260146. eCollection 2023. PMID 37936699
- [Derived] Mao Z, Li X, Korsten K, Bont L, Butler C, Wildenbeest J, Coenen S, Hens N, Bilcke J, Beutels P; RESCEU Investigators. Economic Burden and Health-Related Quality of Life of Respiratory Syncytial Virus and Influenza Infection in European Community-Dwelling Older Adults. J Infect Dis. 2022 Aug 12;226(Suppl 1):S87-S94. doi: 10.1093/infdis/jiac069. PMID 35961055
- [Derived] Zuurbier RP, Korsten K, Verheij TJM, Butler C, Adriaenssens N, Coenen S, Gruselle O, Vantomme V, van Houten MA, Bont LJ, Wildenbeest JG; REspiratory Syncytial Virus Consortium in EUrope (RESCEU) Investigators. Performance Assessment of a Rapid Molecular Respiratory Syncytial Virus Point-of-Care Test: A Prospective Community Study in Older Adults. J Infect Dis. 2022 Aug 12;226(Suppl 1):S63-S70. doi: 10.1093/infdis/jiab600. PMID 35134954
- [Derived] Korsten K, Adriaenssens N, Coenen S, Butler CC, Pircon JY, Verheij TJM, Bont LJ, Wildenbeest JG; RESCEU Investigators. Contact With Young Children Increases the Risk of Respiratory Infection in Older Adults in Europe-the RESCEU Study. J Infect Dis. 2022 Aug 12;226(Suppl 1):S79-S86. doi: 10.1093/infdis/jiab519. PMID 34908153
- [Derived] Korsten K, Adriaenssens N, Coenen S, Butler CC, Verheij TJM, Bont LJ, Wildenbeest JG; RESCEU Investigators. World Health Organization Influenza-Like Illness Underestimates the Burden of Respiratory Syncytial Virus Infection in Community-Dwelling Older Adults. J Infect Dis. 2022 Aug 12;226(Suppl 1):S71-S78. doi: 10.1093/infdis/jiab452. PMID 34904176
- [Derived] Korsten K, Adriaenssens N, Coenen S, Butler C, Ravanfar B, Rutter H, Allen J, Falsey A, Pircon JY, Gruselle O, Pavot V, Vernhes C, Balla-Jhagjhoorsingh S, Oner D, Ispas G, Aerssens J, Shinde V, Verheij T, Bont L, Wildenbeest J; RESCEU investigators. Burden of respiratory syncytial virus infection in community-dwelling older adults in Europe (RESCEU): an international prospective cohort study. Eur Respir J. 2021 Apr 1;57(4):2002688. doi: 10.1183/13993003.02688-2020. Print 2021 Apr. PMID 33060153
- See also: RESCEU consortium webpage — http://resc-eu.org/
- See also: independent multinational research network with the mission to decrease the global burden of RSV infection — http://www.resvinet.org/